CLINICAL TRIAL: NCT02473952
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Immune Globulin (Human), 10% Caprylate/Chromatography Purified (IGIV-C) in Symptomatic Subjects With Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate the Efficacy and Safety of IGIV-C in Symptomatic Subjects With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI1408
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IGIV-C (Experimental): IGIV-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified.
  An initial loading dose of 2 g/kg of body weight will be administered at Baseline (Week 0, Visit 1) followed by maintenance doses of 1 g/kg of body weight administered every third week through Week 21 (Visit 8).
  Interventions: Drug: IGIV-C
- Placebo (Placebo Comparator): Placebo: Sterile 0.9% sodium chloride injection or equivalent. Placebo will be infused at the Baseline/Week 0 Visit (Visit 1) using the same volume as would be required for the IGIV-C loading dose. Subsequent placebo maintenance doses will be matched in volume to the IGIV-C maintenance doses and administered every third week until Week 21 (Visit 8).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IGIV-C — IGIV-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified
  Arms: IGIV-C
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate whether IGIV-C improves MG symptoms as compared to placebo in subjects with MG.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of IGIV-C in subjects with generalized myasthenia gravis (MG) on standard of care treatment at study entry in terms of improvement in MG symptoms as measured by the mean change in Quantitative Myasthenia Gravis (QMG) score from Baseline (Week 0) to Week 24 as compared to placebo.

The safety objective of this study is to evaluate the safety and tolerability of IGIV-C loading dose of 2 g/kg followed by 7 maintenance dosages of 1 g/kg every 3 weeks through Week 21 in subjects with MG.

ELIGIBILITY:
Inclusion Criteria:

* Anti-acetylcholine receptor (AChR) antibody positive
* Confirmed diagnosis of generalized myasthenia gravis (MG).
* Myasthenia Gravis Foundation of America (MGFA) classification of Class II, III, or IVa inclusive at Screening.
* QMG >= 10 at Screening. Note: Subjects who only have a history of ocular MG may not enroll.
* Receiving standard of care MG treatment at a stable dose consisting of any one of the following for the time intervals delineated below (time intervals apply to medications and maintenance of stable dose level):

  1. Cholinesterase inhibitor (pyridostigmine or equivalent) for at least 2 weeks prior to Screening and no immunosuppressants
  2. Cholinesterase inhibitor (pyridostigmine or equivalent) for at least 2 weeks prior to Screening AND/OR only one of the following:

     1. Prednisone (up to 60 mg/day or equivalent) for at least 2 months prior to Screening, OR
     2. Azathioprine for at least 6 months prior to Screening, OR
     3. Mycophenolate mofetil for at least 6 months prior to Screening, OR
     4. Methotrexate for at least 6 months prior to Screening, OR
     5. Cyclosporine or tacrolimus for at least 3 months prior to Screening
  3. Cholinesterase inhibitor (pyridostigmine or equivalent) for at least 2 weeks prior to Screening AND/OR prednisone (up to 60 mg/day or equivalent) for at least one month prior to Screening and only one of the following:

     1. Azathioprine for at least 6 months prior to Screening, OR
     2. Mycophenolate mofetil for at least 6 months prior to Screening, OR
     3. Methotrexate for at least 6 months prior to Screening, OR
     4. Cyclosporine or tacrolimus for at least 3 months prior to Screening

Exclusion Criteria:

* Have received cyclophosphamide or any other immunosuppressive agent apart from the ones allowed per inclusion criteria within the past 6 months
* Any change in MG treatment regimen between Screening (Week -3, Visit 0) and Baseline (Week 0, Visit 1)
* Greater than two point change in QMG score, increased or decreased, between Screening (Week -3, Visit 0) and Baseline (Week 0, Visit 1)
* Any episode of myasthenic crisis in the one month prior to Screening
* Evidence of malignancy within the past 5 years (non-melanoma skin cancer, carcinoma in situ of cervix is allowed) or thymoma potentially requiring surgical intervention during the course of the trial (intent to perform thymectomy)
* Thymectomy within the preceding 6 months
* Rituximab, belimumab, eculizumab or any monoclonal antibody used for immunomodulation within the past 12 months
* Have received immune globulin (Ig) treatment given by intravenous (IV), subcutaneous, or intramuscular route within the last 3 months
* Current known hyperviscosity or hypercoagulable state
* Currently receiving anti-coagulation therapy (vitamin K antagonists, nonvitamin K antagonist oral anticoagulants [e.g., dabigatran etexilate, rivaroxaban, edoxaban, and apixaban], parenteral anticoagulants [e.g., fondaparinux]). Note that oral anti-platelet agents are allowed (e.g., aspirin, clopidogrel, ticlodipine)
* Documented diagnosis of thrombotic complications to polyclonal intravenous immunoglobulin (IVIg) therapy in the past
* History of recent (within the last year) myocardial infarction or stroke
* Uncontrolled congestive heart failure; embolism; or historically documented (within the last year) electrocardiogram (ECG) changes indicative of myocardial ischemia or atrial fibrillation
* History of chronic alcoholism or illicit drug abuse (addiction) in the 12 months preceding the Screening/Week -3 (Visit 0)
* Plasma exchange (PLEX) performed within the last 3 months
* Renal impairment (i.e., serum creatinine exceeds more than 1.5 times the upper limit of normal [ULN] for the expected normal range for the testing laboratory).
* Hemoglobin levels less than 9 g per dL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (15):
  - Phoenix Neurological Associates, Ltd., Phoenix, Arizona
  - University of California-Irvine, Orange, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida Health Science Center, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - London Health Sciences Centre - University Hospital, London, Ontario
  - University Health Network (UHN) - Toronto General Hospital, Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Brno, Dept of Neurologicka klinika, Brno
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
- East Tallinn Central Hospital, Tallinn, Estonia
- France (4):
  - CHU Nice - Hôpital de l'Archet 1, Ctre de Réf Maladies Neuromusculaires et SLA, Nice, Alpes Maritimes
  - CHU Strasbourg - Nouvel Hôpital Civil, Clinique Neurologique, Strasbourg, Bas Rhin
  - CHU de Toulouse - Hôpital Purpan, Service de Neurologie Générale, Toulouse, Haute Garonne
  - Hopital Neurologique Pierre Wertheimer, Neuro-musculaire - Electromyographie, Bron, Rhone
- Germany (7):
  - Universitaetsklinikum Regensburg, Parent, Regensburg, Bavaria
  - Universitaetsmedizin Göttingen, Parent, Göttingen, Lower Saxony
  - Universitaetsklinikum Koeln, Neurologie und Psychiatrie, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Krankenhaus Martha-Maria Halle-Doelau, Klinik fuer Neurologie, Halle, Saxony-Anhalt
  - Universitaetsklinikum Jena, Klinik fuer Neurologie, Jena, Thuringia
  - Universitaetsklinikum Hamburg-Eppendorf, Klinik und Poliklinik fuer Neurologie, Hamburg
- Hungary (3):
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Neurologiai Osztaly, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Neurologia es Stroke Osztaly, Kistarcsa
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Dept of Neurology, Gdansk
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii Klinicznej, Krakow
  - III Szpital Miejski w Lodzi im. Dr K. Jonschera, Lodz
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Dept of Neurology, Warsaw

REFERENCES:
- [Derived] Dalakas MC, Meisel A. Immunomodulatory effects and clinical benefits of intravenous immunoglobulin in myasthenia gravis. Expert Rev Neurother. 2022 Apr;22(4):313-318. doi: 10.1080/14737175.2022.2057223. Epub 2022 Apr 5. PMID 35350948

RESULTS

PARTICIPANT FLOW:
Groups:
- IGIV-C: IGIV-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified.
  An initial loading dose of 2 g/kg of body weight will be administered at Baseline (Week 0, Visit 1) followed by maintenance doses of 1 g/kg of body weight administered every third week through Week 21 (Visit 8).
  IGIV-C: IGIV-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified
- Placebo: Placebo: Sterile 0.9% sodium chloride injection or equivalent. Placebo will be infused at the Baseline/Week 0 Visit (Visit 1) using the same volume as would be required for the IGIV-C loading dose. Subsequent placebo maintenance doses will be matched in volume to the IGIV-C maintenance doses and administered every third week until Week 21 (Visit 8).
  Placebo
Period: Overall Study
Arm/Group | IGIV-C | Placebo
Started | 30 | 32
Completed | 28 | 24
Not Completed | 2 | 8
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV-C | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (17.06) | 48.0 (13.66) | 51.2 (15.63)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 20 | 29 | 49
  >=65 | 10 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 11 | 12 | 23
  Europe | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Myasthenia Gravis (MG) Symptoms as Measured by the Mean Change in Quantitative Myasthenia Gravis (QMG) Total Score.
Description: To measure improvement in MG symptoms by the mean change in QMG total score from Baseline (Week 0) to Week 24 as compared to placebo. Evaluators score 13 individual items (range from 0=best to 3=worst) and the individual scores are added together for the total score (range 0-39). An average 3-point improvement in QMG score indicates clinically meaningful improvement.
Time Frame: Baseline (Week 0) to Week 24
Population: Modified intent-to-treat population consisting of all randomized subjects who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | -4.6 (5.11) | -2.7 (6.23)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from screening through Week 24.
Arm/Group | IGIV-C | Placebo
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 5/30 | 4/32
Other Adverse Events (participants affected / at risk) | 22/30 | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C (N=30) | Placebo (N=32)
Myasthenia gravis (Nervous system disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C (N=30) | Placebo (N=32)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (13) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 9 (22) | 4 (6)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 2 (2)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 3 (5) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing Sponsor at least thirty days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At Sponsor's request, the site will remove any confidential information (other than study results), and incorporate all reasonable comments by Sponsor, or delay publication or presentation for a period of up to 120 days to allow Sponsor to protect its interests in any Sponsor's Inventions.

DOCUMENTS (2):
  • Study Protocol (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT02473952/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT02473952/SAP_001.pdf